CLINICAL TRIAL: NCT01129323
Title: Reduced-Intensity Preparative Regimen for Allogeneic Stem Cell Transplantation in Patients With Severe Aplastic Anemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study did not accrue any subjects and due to this will be closed.
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07081
Record Dates: First submitted 2010-04-21; First posted 2010-05-24 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Severe Aplastic Anemia
Keywords: Anemia, Severe, Aplastic, Reduced-Intensity, Allogeneic, Stem, Cell, Transplantation
MeSH Terms: conditions — Anemia, Aplastic; Anemia | interventions — Cyclophosphamide; fludarabine; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reduced-Intensity Preparative Regimen for Allogeneic SCT (Experimental): Patient in this arm will receive maximally tolerated (reduced) doses of cytotoxic therapy with the goals of suppressing the immune system, and ablate host hematopoiesis to ensure engraftment of the donor's hematopoietic system.
  Interventions: Drug: Cyclophosphamide, Fludarabine, Rabbit ATG

INTERVENTIONS:
Drug: Cyclophosphamide, Fludarabine, Rabbit ATG — Fludarabine 30mg/m2/dose IV and cyclophosphamide 10mg/kg/dose IV are given once per day from day -5 to -2. rATG 1.5 mg/kg/dose IV is given from day -4 to -1.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of allogeneic transplant after a reduced-intensity preparative regimen for patient, to evaluate survival, and to evaluate the side effects of this treatment. The patient will be in the study for two years for treatment and active monitoring. After treatment and active monitoring are over, the patient's medical condition will be followed indefinitely.

DETAILED DESCRIPTION:
Aplastic Anemia is a blood disorder where bone marrow does not produce enough cells for blood. Patients with aplastic anemia have lower counts of all three blood cell types (RBC, WBC, and Platelet). Severe cases of aplastic anemia that are untreated can lead to death from bleeding and overwhelming infection.

For patients with Severe Aplastic Anemia (SAA), allogeneic hematopoietic stem cell transplant (HSCT) from an HLA-identical sibling is an accepted treatment for restoring normal bone marrow function. Preparative regimens for allogeneic HSCT are designed to give the highest tolerated doses of chemotherapy, with or without total body irradiation (TBI), in order to fully "ablate" or destroy the patient host's bone marrow so that the transplanted cells from the HLA-identical sibling can engraft in the patient host.

While allogeneic HSCT has been proven to be a curative form of therapy for SAA, it is also associated with high transplant-related morbidity (side effects) and possible mortality (death). One of the toxic side effects from high-dose chemotherapy and TBI are believed to be a major contributing factor to "Graft-versus-Host Disease" (GVHD).

Preliminary studies have shown that a reduced intensity (non-myeloablative) allogeneic HSCT may be just as effective in treating SAA. Low-dose chemotherapy is used instead of high-dose chemotherapy and TBI. Some smaller studies have indicated that reduced intensity preparative regimens using Fludarabine and Cyclophosphamide allowed engraftment in the matched sibling donor setting with an acceptable level of toxic side effects in subjects with a variety of hematologic cancers. Additional studies that followed showed that a reduced intensity preparative regimen that included fludarabine, cyclophosphamide and antithymocyte globulin, allowed engraftment of donor stem cells in subjects with SAA with acceptable engraftment rates and a decrease in the severity of GVHD.

This study is designed to evaluate the effectiveness of allogeneic transplant after a reduced-intensity preparative regimen, to evaluate survival, and to evaluate the side effects including GVHD of this treatment. Patients will be in the study for two years for treatment and active monitoring. All patients will be followed until death.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or younger
* Male or female recipients must have histopathologically confirmed diagnosis of severe aplastic anemia. Diagnostic Criteria for Server Aplastic Anemia will be based on the definitions set forth by the international Aplastic Anemia Study Group
* At least two of the following:

Absolute neutrophil count <0.5 x 109/L Platelet count <20 x 109 /L Anemia with corrected reticulocyte count <1%

AND

* Bone marrow cellularity <25%, or bone marrow cellularity <50% with fewer than 30% hematopoietic cell
* Availability of an HLA identical sibling

Exclusion Criteria:

* Active and uncontrolled infection
* HIV-1 infection
* Pregnancy or breastfeeding.
* DLCO <40% predicted
* Left Ventricular Ejection Fraction < 40%
* Performance scale Karnofsky <=40% or Lansky<=40% for patients <16 years old

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Engraftment rate | Day 42 after allogeneic transplant

SECONDARY OUTCOMES:
Relapse | Days 180, 365 and yearly post transplant
Development of Graft vs. Host Disease | Days 180, 365 and yearly post transplant
Evaluation of the occurrence of secondary malignancies | Days 180, 365 and yearly post transplant
Overall survival | Days 180, 365 and yearly post transplant
Evaluation of treatment feasibility | Days 180, 365 and yearly post transplant
Evaluation of toxicities | Days 180, 365 and yearly post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pawlowska, MD, Principal Investigator — City of Hope Medical Center